CLINICAL TRIAL: NCT02693249
Title: Dysfunctional Posttraumatic Cognitions in Children and Adolescents
Acronym: PTC
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016-00275
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-03

CONDITIONS: Motor Vehicle Accident; Burns
Keywords: accidents; adolescents; children; posttraumatic cognitions
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the psychological consequences of motor vehicle accidents and burn accidents in 7-18 years old children and adolescents. The impact of posttraumatic cognitions on developing psychological symptoms are of particular interest.

DETAILED DESCRIPTION:
Background: Dysfunctional trauma-related cognitions play an important role in the aftermath of a traumatic event. Children and adolescents, who think that the experienced trauma has a permanent and disturbing impact on their actual life and their future, feel threatened. Study results show that dysfunctional posttraumatic cognitions correlate highly with posttraumatic stress symptoms (PTSS), depression, and anxiety. In addition, children and adolescents with a posttraumatic stress disorder (PTSD) have significantly more dysfunctional trauma-related cognitions than those without PTSD. Especially for children and adolescents it is important to consider interacting developmental and environmental factors. A developmental approach, nevertheless, has not been investigated yet.

Aims: The aims of the proposed study are to achieve a better understanding of dysfunctional trauma-related cognitions considering child and environmental factors in a cross-sectional and a longitudinal design.

Method: The sample consists of two different subsamples: 1) A hospital sample consisting of children and adolescents (school age: 7-18 years), who experienced an accidental trauma (either acute traffic accident or burn injury) assessed at three times: in the acute phase (7-14 days), 3 months, and 6 months after the trauma occurred. 2) An already existing clinical sample of 159 children and adolescents (TreatChildTrauma study), who mostly experienced an interpersonal trauma such as sexual or physical abuse. The total sample will be used to investigate the impact of child and environmental factors including trauma type, trauma frequency, age, gender, risk status pre trauma (psychopathological status pre trauma and traumatic events pre trauma), psychopathological status post trauma, and parental trauma-related cognitions. In addition, the hospital sample will be used for assessing the naturalistic time course of dysfunctional trauma-related cognitions as well as the association between cognitions, PTSS, depression, and anxiety over time. Moreover, the association between parental dysfunctional trauma-related cognitions and altered parenting as well as their impact on the child's cognitions will be investigated.

Relevance: Dysfunctional trauma-related cognitions have an important impact on coping with a traumatic event in childhood and adolescence. Nevertheless, no study has investigated the interaction between several child and environmental factors so far. A gain of knowledge in this area is important to improve treatments of trauma-related disorders.

ELIGIBILITY:
Inclusion Criteria:

* child age between 7.0 and 18.0
* outpatient or inpatient medical care at the University Children's Hospital Zurich because of an injury after a traffic accident or a burn accident
* at least one parent participating

Exclusion Criteria:

* a severe comorbid head injury (Glasgow Coma Scale < 9)
* any previous evidence of pervasive developmental disorder
* an insufficient command of the German language of the participant or of the parents

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents (ages 7-18 years), who experienced an accidental trauma (either traffic accident or burn accident) and at least one parent.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Child Posttraumatic Cognitions Inventory (CPTCI) | 6 months
  The CPTCI is a 25-item self-report measure assessing dysfunctional posttraumatic cognitions in children ages 6-18 years. The questionnaire showing good psychometric properties yields scores for two subscales "Permanent and disturbing change" and "Fragile person in a scary world" as well as a total score.

SECONDARY OUTCOMES:
University of California at Los Angeles Post-Traumatic Stress Disorder Reaction Index DSM-5 version (UCLA PTSD RI DSM-5) | 6 months
  The UCLA PTSD RI DSM-5 is a widely used and well validated questionnaire assessing posttraumatic stress symptoms in children and adolescents ages 7-18 years. Both self-report and proxy-report will be used.
Children's Depression Inventory (CDI) | 6 months
  The CDI is a 29-item self-report measure assessing depression symptoms in children ages 8-16 years. The questionnaire showing good psychometric properties yields a total score.
Screen for Child Anxiety Related Disorders (SCARED) | 6 months
  The SCARED is a 41-item self-report measure assessing anxiety symptoms in children ages 8-18 years which shows good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Markus A. Landolt, Prof. Dr., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No